CLINICAL TRIAL: NCT00055887
Title: A Phase III Randomized, Open-Label Comparative Study of Induction Chemotherapy Followed by Thoracic Radiation Therapy With Supplemental Oxygen, With or Without Concurrent RSR13 (Efaproxiral), in Patients With Locally Advanced Unresectable (Stage IIIA/IIIB) Non-Small Cell Lung Cancer
Brief Title: Chemotherapy and Radiation Therapy With or Without Efaproxiral in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never started. No patients were enrolled.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000271438; ALLOS-RSR13RT-013ELITE
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IIIA non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Cisplatin; efaproxiral; Gemcitabine; Paclitaxel; Vinorelbine; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: efaproxiral
Drug: gemcitabine hydrochloride
Drug: paclitaxel
Drug: vinorelbine ditartrate
Procedure: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as efaproxiral may make the tumor cells more sensitive to radiation therapy. It is not yet known if chemotherapy combined with radiation therapy is more effective with or without efaproxiral in treating non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy combined with radiation therapy with or without efaproxiral in treating patients who have stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with stage IIIA or IIIB non-small cell lung cancer treated with induction chemotherapy followed by radiotherapy with or without efaproxiral.
* Compare time to progression, response rate, and pattern of failure of patients treated with these regimens.
* Determine the safety of efaproxiral in these patients.
* Determine the pharmacokinetics of efaproxiral in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to chemotherapy regimen, Karnofsky performance status (70-80% vs 90-100%), and disease stage (IIIA vs IIIB).

* Induction therapy phase: Patients receive 1 of the following induction chemotherapy regimens:

  * Paclitaxel and carboplatin: Patients receive paclitaxel IV and carboplatin IV on day 1. Treatment repeats every 21 days for a total of 2 courses.
  * Cisplatin and gemcitabine: Patients receive cisplatin IV on day 2 and gemcitabine IV on days 1, 8, and 15. Treatment repeats every 28 days for a total of 2 courses.
  * Cisplatin and vinorelbine: Patients receive cisplatin IV on day 1 and vinorelbine IV on days 1, 8, and either 15 or 22. Treatment repeats every 28 days for a total of 2 courses.
* Randomized phase: Within 42 days after completion of chemotherapy, patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive efaproxiral IV over 30-45 minutes with supplemental oxygen and then undergo concurrent radiotherapy 5 days a week for 7 weeks.
  * Arm II: Patients receive supplemental oxygen and undergo radiotherapy as in arm I.

Quality of life is assessed at baseline, on days 1 and 16 of radiotherapy, monthly for 3 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

Patients are followed monthly for 3 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 659 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced, unresectable non-small cell lung cancer of 1 of the following subtypes:

  * Adenocarcinoma
  * Squamous cell carcinoma
  * Large cell carcinoma
  * Poorly differentiated carcinoma
* Stage IIIA or IIIB

  * T1 or T2, N2
  * T3, N1 or N2
  * T4, any N
  * Any T, N3
* Histological or cytological confirmation of at least 1 positive lymph node required if the largest mediastinal node that is the basis of stage III disease is less than 2.0 cm in diameter
* Clinically or radiologically measurable disease of at least 2.0 cm
* Partially resected stage IIIB disease allowed provided a measurable lesion remains
* No pleural effusion that is bloody, cytologically positive, or re-accumulated after thoracentesis
* No metastatic disease by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin at least 10 g/dL
* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No clinically active congestive heart failure
* No unstable angina
* No severe arrhythmia by ECG

Pulmonary

* FVC and FEV_1 at least 50% of normal
* Resting oxygen saturation by pulse oximetry (SpO_2) at least 90% on room air
* Exercise SpO_2 at least 90% on room air

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective contraception during and for 30 days after study therapy
* Male patients must use effective contraception during and for 90 days after study therapy
* No loss of more than 10% of body weight within the past 3 months
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No significantly altered mental status or dementia that would preclude giving informed consent
* No active infection
* No other serious underlying medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy
* No concurrent colony-stimulating factors (randomized phase only)
* No biologic therapy during and for 1 month after study therapy
* No immune response modifiers during and for 1 month after study therapy

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* No hormonal therapy during and for 1 month after study therapy

Radiotherapy

* No prior thoracic radiotherapy

Surgery

* See Disease Characteristics
* No prior total surgical resection

Other

* More than 28 days since prior investigational drugs or devices
* No prior efaproxiral
* No other cytotoxic therapy during and for 1 month after study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-11

CONTACTS AND LOCATIONS:
Overall Officials: Hak Choy, MD, Study Chair — Simmons Cancer Center
Locations (22):
- United States (8):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Cancer Center at Lexington Clinic, Lexington, Kentucky
  - Willis - Knighton Cancer Center, Shreveport, Louisiana
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Providence Everett Medical Center - Pacific Campus, Everett, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
- Algemeen Ziekenhuis Middelheim, Antwerp, Belgium
- Canada (9):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Notre- Dame du CHUM, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky